CLINICAL TRIAL: NCT01715181
Title: A Cluster-Randomized Controlled Trial Evaluating the Effects of a Volunteer-Led Nonpharmacological Intervention to Reduce Neuropsychiatric Symptoms of Dementia in Long-Term Care Residents
Brief Title: Volunteers Adding Life in Dementia: VALID
Acronym: VALID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Dr. Dallas Seitz, Assistant Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VALIDII; NIRG-12-236827 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Individuals will receive usual care
- Volunteer visits (Experimental): Volunteers will visit 3 times per week with a visit duration of 30 minutes for each visit during the study.
  Interventions: Other: Volunteer visits

INTERVENTIONS:
Other: Volunteer visits — Volunteers will visit 3 times per week with a visit duration of 30 minutes for each visit during the study.
  Arms: Volunteer visits

SUMMARY:
Older adults with Alzheimer's disease and other forms of dementia frequently develop challenging neuropsychiatric symptoms (NPS) as a result of their illness. Non-pharmacological strategies to manage these symptoms such as music, exercise, and participating in pleasant social events have been demonstrated to be safe and effective strategies to reduce these behavioral symptoms. Our project, Volunteers Adding Life in Dementia (VALID), will design and implement a volunteer-led program to reduce behavioral symptoms and improve the quality of life of older adults with dementia who are residing in long-term care facilities.

DETAILED DESCRIPTION:
The number of older adults with Alzheimer's disease (AD) and related forms of dementia is increasing in Canada and the majority of individuals with dementia develop neuropsychiatric symptoms (NPS) such as agitation, psychosis, depression and anxiety at some time during their illness. NPS are particularly problematic in long-term care (LTC) where approximately 60% of individuals have dementia, and 80% of individuals with dementia have NPS at any time. Adverse outcomes associated with NPS include increased use of psychotropic medications, stress for families and nursing staff, increased costs of care, and decreased quality of life. A novel approach to implementing non-pharmacological interventions for LTC residents with NPS is the use of volunteers. Volunteer-led programs have been demonstrated to be an effective, inexpensive, and sustainable method of implementing psychosocial interventions for older adults in acute care. The objectives of our project are to: 1.) Recruit and train approximately 40 volunteers in the VALID program; 2.) Conduct a cluster-randomized controlled trial of the VALID program in 6 LTC facilities (3 intervention and 3 control LTC sites; 60 individuals with dementia in each of the experimental and control arms) to determine the effect of the VALID program on symptoms of NPS, patient quality of life, volunteer's experience, and LTC staff stress, 3.) Determine key components of the VALID program that served as facilitators and barriers to implementation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Alzheimer's disease or related forms of dementia
* significant symptoms of agitation as measured by a Cohen-Mansfield Agitation Inventory (CMAI) total score of >39
* resident in LTC facility for at least 30 days
* presence of a caregiver or substitute decision maker willing to consent to treatment
* no changes in psychotropic medications in the 2 weeks preceding enrolment in study

Exclusion Criteria:

* depressive symptoms presenting acute risk (i.e. suicidal ideation)
* physically aggressive behavior posing safety risk to others
* uncontrolled pain
* currently receiving palliative care
* medically unstable with life expectancy of < 6 months
* currently awaiting transfer to another LTC facility or hospital

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in neuropsychiatric symptoms (measured by the Cohen-Mansfield Agitation Inventory) | Baseline, weeks 2,4,6,8 and 12

SECONDARY OUTCOMES:
Change in Neuropsychiatric Inventory score | Baseline, weeks 4, 8, 12
Change in Cornell Depression in Dementia Rating Scale score | Baseline, weeks 4, 8, 12
Change in Dementia Quality of Life Scale (DEMQoL) score | Baseline, weeks 4, 8, 12
Change in Clinical Global Impression of Change (CGI-C)score | 12 weeks

OTHER OUTCOMES:
Modified nursing care assessment scale (M-NACS) | Baseline, week 12
Short Form Health Survey | Baseline, week 12
  Assessment of volunteer quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dallas P Seitz, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada